CLINICAL TRIAL: NCT03367130
Title: Integrating Mobile Phone-Based Intervention With Test and Treat Strategy to Improve Clinic Attendance for Antiretroviral Pills Pick Up Among HIV Positive Individuals in Nepal: A Randomized Controlled Trial
Brief Title: Improving Clinic Attendance for Medication Collection Among HIV Positive Individuals in Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo University (Other)
Collaborators: Asian Development Bank Japan Scholarship Program (Unknown); Open Society Institute (Unknown)
Responsible Party: Principal Investigator, Rakesh Ayer, Mr., Tokyo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 11711
Record Dates: First submitted 2017-12-03; First posted 2017-12-08 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: HIV Infections; Antiretroviral Therapy; HIV Seropositivity
Keywords: Antiretroviral therapy, clinic attendance, Nepal
MeSH Terms: conditions — HIV Infections; HIV Seropositivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This study will be a double blinded RCT. HIV-positive individuals will be blinded to allocation group. Further, those who deliver the intervention will be blinded to the allocation. Intervention and control groups will receive similar intervention strategies. Only the content of the interventions will be different. Therefore, it is difficult for HIV-positive individuals to tell if they are receiving intervention or control. The outcome assessor will be masked to the allocation of each HIV-positive individual by using trial identity numbers. Only the principal researcher will have complete access to all the information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): HIV-positive individuals will receive the standard HIV care following the national ART guidelines. In addition, the intervention group will receive mobile phone calls. A mobile phone reminder will be made two days prior to their scheduled appointment for pills pick up. Trained research assistants will remind them of their scheduled clinic appointment of pills pick up. If the first call is missed, the second call will be made within the same day, if the second call is also missed, the final call will be made next day. The intervention will be delivered over the period of six months. Outcome assessors will not be involved in the phone calls.
  Interventions: Behavioral: Mobile phone reminder
- Control (Placebo Comparator): Control group will also receive the standard HIV care following the national ART guidelines and phone calls educating them on healthy living. Phone calls will be made once a month.
  Interventions: Behavioral: Mobile phone reminder

INTERVENTIONS:
Behavioral: Mobile phone reminder — Intervention described already in arm/group descriptions.

SUMMARY:
Antiretroviral therapy (ART) has been a game changer in the context of HIV-epidemic. From 2005 to 2015, HIV-related deaths have fallen by 45% thanks to ART. However, ART's success heavily depends on HIV-positive individuals' high adherence to it. This includes clinic attendance for various purposes. It is necessary among HIV-positive individuals for their antiretroviral (ARV) pills pick up, monitoring of their treatment outcomes, and treatment of their opportunistic infections. Among them, ARV pills pick up is the major reason for the ART clinic attendance. Improving clinic attendance for pills pick up remains one of the key challenges to ART programs. The World Health Organization (WHO) recommends more than 90% on-time ARV pills pick up as per the early warning indicators of HIV-drug resistance. Among six Asian countries, none of the 1048 clinics under the study could meet the WHO target. Among HIV-positive individuals, clinic attendance for pills pick can be improved by using mobile phones. Those who receive mobile phone reminders are two times more likely to attend their clinics regularly than those who did not receive such reminders. Nepal belongs to a low-income country and is facing a similar problem, too. In 2015, approximately 39,000 people were estimated to be living with HIV and ART coverage was limited to only 31.5%. In the same year, only 32% of the HIV-positive individuals attended their clinics regularly for ARV pills pick up. Like other countries, one of the potential strategies is to use mobile phones effectively in Nepal. Mobile phones have been very widely used in Nepal. In 2016, Nepal had 27.9 million mobile phone users, against the population of 26.5 million. Under such a context, mobile phone reminders can be effective to improve clinic attendance among HIV-positive individuals. However, the effectiveness of such interventions barely remains examined by using a randomized controlled trial. This study evaluates the effectiveness of mobile phone reminder intervention on improving clinic attendance for ARV pills pick up and medication adherence among HIV-positive individuals on ART following the implementation of test and treat strategy in Nepal.

DETAILED DESCRIPTION:
Background Antiretroviral therapy (ART) has been a game changer in the context of HIV-epidemic. From 2005 to 2015, HIV-related deaths have fallen by 45% thanks to ART. In addition, ART has produced a two-fold positive impact on the lives of HIV-positive populations. First, it has increased the life expectancy and improved the quality of life of HIV-positive individuals. Second, it has prevented new infections in the population.

However, ART's success heavily depends on HIV-positive individuals' high adherence to it. This includes clinic attendance for various purposes. It is necessary among HIV-positive individuals for their antiretroviral (ARV) pills pick up, monitoring of their treatment outcomes, and treatment of their opportunistic infections. Among them, ARV pills pick up is the major reason for the ART clinic attendance.

Three negative consequences may occur when HIV-positive individuals miss their clinic attendances. First, it can directly impair their medication adherence. Second, HIV-drug resistance and treatment failure could rise. Finally, mortality may increase among HIV-positive individuals. In addition, missed clinic attendances increase economic burden to the health system. However, both in high-and low-income countries, significant proportions of HIV-positive individuals miss their scheduled clinic attendances for ARV pills pick up.

Improving clinic attendance for pills pick up remains one of the key challenges to ART programs. The World Health Organization (WHO) recommends more than 90% on-time ARV pills pick up as per the early warning indicators of HIV-drug resistance. However, in 2012, worldwide, more than 30% of the ART clinics did not meet WHO target of timely ARV pills pick up.

Achieving WHO's pills pick up target is more challenging in low-income countries. For instance, in the Sub-Saharan Africa, 59 to 83% of the ART clinics could not achieve the WHO target of on-time pills pick up. Similarly, among six Asian countries, none of the 1048 clinics under the study could meet the WHO target.

Among HIV-positive individuals, clinic attendance for pills pick can be improved by using mobile phones. Mobile phones are generally used in two ways. First, a voice call is used to remind HIV-positive individuals about their scheduled clinical appointments. Second, a short message is sent to HIV-positive individuals to remind them about their appointments. Those who receive mobile phone reminders are two times more likely to attend their clinics regularly than those who did not receive such reminders. Particularly, mobile phone reminders have shown positive effects to improve clinic attendance for pills pick up in low-income settings.

Nepal belongs to a low-income country and is facing a similar problem, too. In 2015, approximately 39,000 people were estimated to be living with HIV, and ART coverage was limited to only 31.5% of the total eligible people. In the same year, only 32% of the HIV-positive individuals attended their clinics regularly for ARV pills pick up. They faced barriers to regular clinic attendance such as a dearth of family support, long commuting time, lack of ART knowledge, and non-participation in support programs.

To improve the HIV-positive individuals' health status, the Government of Nepal (GoN) has made significant decisions at the national level. Free ART services were the primal ones. It consists of free ARV drugs and care package including follow-up, tuberculosis screening, isoniazid preventive therapy, community and home-based care. GoN initiated the free ART service in 2004 from Sukra Raj Tropical and Infectious Disease Control Hospital, Teku, Kathmandu. Since the first initiation, the ART services have been provided through more than 60 ART clinics located in non-governmental and government health facilities. From 2017, Nepal has also started a test and treat strategy recommended by WHO to achieve 90-90-90 targets by 2020 and ending AIDS epidemic by 2030. However, limited efforts have been made to improve ARV pills pick up. Therefore, effective strategies are urgently needed to improve on-time ARV pills pick up.

Like other countries, one of the potential strategies is to use mobile phones effectively in Nepal. Mobile phones have been very widely used since the beginning of 21st century, and its coverage has exceeded 100% compared to the total population. In 2016, Nepal had 27.9 million mobile phone users, against the population of 26.5 million. Under such a context, mobile phone reminders can be effective to improve clinic attendance among HIV-positive individuals. However, the effectiveness of such interventions barely remains examined by using a randomized controlled trial. This study evaluates the effectiveness of mobile phone reminder intervention on improving clinic attendance for ARV pills pick up and medication adherence among HIV-positive individuals on ART after the implementation of test and treat strategy in Nepal.

Methods Study design This study is a two-arm randomized controlled trial with an HIV-positive person as the unit of randomization. The allocation ratio will be 1:1.

Sample and Setting In 2016, 63 ART clinics were functional in Nepal. Out of 63 clinics, 18 clinics have a CD4 cell testing facility. As of May 2017, about 12,000 HIV positive individuals were accessing these services. This study will be conducted at public ART clinics in Kathmandu, Rupandehi, Banke, Kailali, and Kanchanpur districts of Nepal.

All the study clinics are under the Nepalese Ministry of Health. According to the information from all of these target ART clinics, about 7000 HIV-positive individuals were accessing ART services by May 2017.

This study will be carried from November 2017 to May 2018. These HIV-positive individuals will be followed up for six months.

Sample size Clinic attendance is the primary outcome variable in this study. Based on the previous study, I assumed regular clinic attendance rate of 33%. If the intervention increased the rate from 33% to 48% (approximately 15 percentage points), then about 370 HIV-positive individuals, 185 in the intervention and 185 in the control group, would be required to reject the null hypothesis that no difference exists between intervention and the control group at the end of the follow up period. To counter for lost to follow-up and missing data, I will recruit 600 HIV-positive individuals in total (intervention: 300 and control: 300). I also assumed 95% confidence interval and 80% power of the test.

Enrolment procedure At first, the eligibility criteria will be assessed based on the medical records, and all the eligible HIV-positive individuals will be invited to participate in the trial. Next, written consent will be sought from each HIV-positive individual and then they will be enrolled in the study. Enrollment will take place at each ART clinic.

Randomization and allocation concealment ART numbers are known as patient identification numbers for HIV-positive individuals and they will be used in this study to maintain anonymity. Trial assistants will collect the ART numbers of HIV-positive individuals. In this study, their ART numbers will be converted to unique trial identity numbers to maintain the confidentiality in the trial. An independent researcher will randomize the trial identity numbers after collecting the background information. HIV-positive individuals will be randomized to either the intervention group or the control group using a computer random number generator (1:1 randomization).

Blinding This study will be a double-blinded RCT. HIV-positive individuals will be blinded to allocation group. Further, those who deliver the intervention will be blinded to the allocation.

Intervention and control groups will receive similar intervention strategies. Only the content of the interventions will be different. Therefore, it is difficult for HIV-positive individuals to tell if they are receiving intervention or control. The outcome assessor will be masked to the allocation of each HIV-positive individual by using trial identity numbers. Only the principal researcher will have complete access to all the information.

Interventions

Intervention arm:

HIV-positive individuals will receive the standard HIV care following the national ART guidelines. In addition, the intervention group will receive mobile phone calls. A mobile phone reminder will be made two days prior to their scheduled appointment for pills pick up. Trained research assistants will remind them of their scheduled clinic appointment of pills pick up. If the first call is missed, the second call will be made within the same day, if the second call is also missed, the final call will be made next day. The intervention will be delivered over the period of six months. Outcome assessors will not be involved in the phone calls.

Control arm:

Control group will also receive the standard HIV care following the national ART guidelines and phone calls educating them on healthy living. Phone calls will be made once a month.

Withdrawal from study HIV-positive individuals will be given full right to withdraw from this trial at any stage. However, reasons for their withdrawal will be sought from them and will be appropriately recorded.

A mixed-method (cross-sectional study and in-depth interviews) study will be conducted prior to the intervention.

Outcome assessment Outcome data will be obtained from the medical records of HIV-positive individuals maintained at the ART clinics. ART medication adherence data will be collected by telephone interview. I will measure the effect of a mobile phone reminder intervention on clinic attendance and medication adherence using generalized estimating equation. An interviewer-administered, pre-tested questionnaire would be used to collect the data.

Trained research assistants will assess and collect data related to outcome in the coded form. These research assistants will not be involved in the intervention delivery. Collected data will be entered in EpiData software version 3.1(EpiData Association Denmark).

I will conduct a training on data collection for research assistants. The training includes ethical issues, data collection and communication with HIV-positive individuals.

Data analyses The background characteristics of HIV-positive individuals will be compared between intervention and control group using the chi-squared test or Fisher's exact test. These tests will be used to compare the proportions, and Student's t-test will be used to compare means. Main data analyses will be conducted on intention-to-treat principle. A relevant multiple imputation method will be applied for completely missing data related to primary and secondary outcomes. HIV-positive individuals' retention in trial will be measured by an instrumental variable method. I will perform all analysis with two-sided tests with a 5% level of significance. STATA software version 13.1(College Station, Texas, USA) will be used for data analyses.

Ethical Consideration Ethical approval will be first sought from the Research Ethics Committee of the University of Tokyo and Nepal Health Research Council, Nepal. In addition, written approval will be obtained from each study hospital. Written informed consent will all be sought from each HIV-positive individual.

HIV-positive individuals will be given full right to withdraw from this trial at any stage of the intervention. However, reasons for their withdrawal will be sought from them and will be appropriately recorded.

ELIGIBILITY:
Inclusion criteria

* Eligibility criteria

  1. be 18 years or over;
  2. own a mobile phone;
  3. started treatment following test and treat strategy; and
  4. under the first line ART regimen
* Exclusion criteria HIV-positive individuals will be excluded if they have severe physical and mental illnesses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2017-10-14 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Clinic attendance for pills pick up | six months.
  Clinic attendance adherence rate will be used to assess the clinic attendance. The rate will be based on the rate of total days adhered to the total scheduled days. An attendance will be called 'adhered', when they maintained an attendance in less than or equals to two days among scheduled days. Information on clinic attendance will be obtained from HIV-positive individuals' treatment and care files. Clinic attendance will be measured over the period of six months after the intervention.
  Dichotomous measure will be used to assess the clinic attendance for pills pick up. A 100% adherence rate will be used to define regular clinic attendance and missing any appointment(s) will be categorized as inconsistent clinic attendance.

SECONDARY OUTCOMES:
Delay in pills pick up | Six months.
  Delay in pills pick up will be assessed with the number of days late from the scheduled appointment to the actual date of medication collection.
Medication adherence | Six months.
  Medication adherence will be measured at the baseline and at the end of the intervention. The questionnaire will be adopted from AIDS Clinical Trials Group. Intake of >95% of the doses of prescribed will be defined as adherent and intake of <= 95% of the doses will be defined as non-adherent. Possible reasons will also be collected for missing to take medications.

CONTACTS AND LOCATIONS:
Overall Officials: Masamine Jimba, PhD, MD, MPH, Study Chair — Tokyo University
Locations (1):
- Seti Zonal Hospital, Dhangadi, State 7., Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Medland NA, McMahon JH, Chow EP, Elliott JH, Hoy JF, Fairley CK. The HIV care cascade: a systematic review of data sources, methodology and comparability. J Int AIDS Soc. 2015 Nov 30;18(1):20634. doi: 10.7448/IAS.18.1.20634. eCollection 2015. PMID 26626715
- [Background] Havlir D, Beyrer C. The beginning of the end of AIDS? N Engl J Med. 2012 Aug 23;367(8):685-7. doi: 10.1056/NEJMp1207138. Epub 2012 Jul 18. No abstract available. PMID 22809362
- [Background] Cohen MS, Smith MK, Muessig KE, Hallett TB, Powers KA, Kashuba AD. Antiretroviral treatment of HIV-1 prevents transmission of HIV-1: where do we go from here? Lancet. 2013 Nov 2;382(9903):1515-24. doi: 10.1016/S0140-6736(13)61998-4. Epub 2013 Oct 23. PMID 24152938
- [Background] UNAIDS. Global AIDS update 2016. Geneva, Switzerland: Joint United Nations Programme on HIV/AIDS; 2016.
- [Background] Byass P. Cause-specific mortality findings from the Global Burden of Disease project and the INDEPTH Network. Lancet Glob Health. 2016 Nov;4(11):e785-e786. doi: 10.1016/S2214-109X(16)30203-0. No abstract available. PMID 27765285
- [Background] Consolidated Guidelines on the Use of Antiretroviral Drugs for Treating and Preventing HIV Infection: Recommendations for a Public Health Approach. 2nd edition. Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK374294/ PMID 27466667
- [Background] Shumba C, Atuhaire L, Imakit R, Atukunda R, Memiah P. Missed Doses and Missed Appointments: Adherence to ART among Adult Patients in Uganda. ISRN AIDS. 2013 Jan 14;2013:270914. doi: 10.1155/2013/270914. eCollection 2013. PMID 24052886
- [Background] WHO. World health organization global strategy for the surveillance and monitoring of HIV drug resistance. Geneva, Switzerland: World Health Organization, 2012.
- [Background] Perron NJ, Dao MD, Kossovsky MP, Miserez V, Chuard C, Calmy A, Gaspoz JM. Reduction of missed appointments at an urban primary care clinic: a randomised controlled study. BMC Fam Pract. 2010 Oct 25;11:79. doi: 10.1186/1471-2296-11-79. PMID 20973950
- [Background] Bennett DE, Jordan MR, Bertagnolio S, Hong SY, Ravasi G, McMahon JH, Saadani A, Kelley KF. HIV drug resistance early warning indicators in cohorts of individuals starting antiretroviral therapy between 2004 and 2009: World Health Organization global report from 50 countries. Clin Infect Dis. 2012 May;54 Suppl 4(Suppl 4):S280-9. doi: 10.1093/cid/cis207. PMID 22544188
- [Background] Fokam J, Billong SC, Bissek AC, Kembou E, Milenge P, Abessouguie I, Nkwescheu AS, Tsomo Z, Aghokeng AF, Ngute GD, Ndumbe PM, Colizzi V, Elat JB. Declining trends in early warning indicators for HIV drug resistance in Cameroon from 2008-2010: lessons and challenges for low-resource settings. BMC Public Health. 2013 Apr 8;13:308. doi: 10.1186/1471-2458-13-308. PMID 23565992
- [Background] Kunutsor S, Walley J, Katabira E, Muchuro S, Balidawa H, Namagala E, Ikoona E. Using mobile phones to improve clinic attendance amongst an antiretroviral treatment cohort in rural Uganda: a cross-sectional and prospective study. AIDS Behav. 2010 Dec;14(6):1347-52. doi: 10.1007/s10461-010-9780-2. PMID 20700644
- [Background] Abdulrahman SA, Rampal L, Ibrahim F, Radhakrishnan AP, Kadir Shahar H, Othman N. Mobile phone reminders and peer counseling improve adherence and treatment outcomes of patients on ART in Malaysia: A randomized clinical trial. PLoS One. 2017 May 16;12(5):e0177698. doi: 10.1371/journal.pone.0177698. eCollection 2017. PMID 28520768
- [Background] Free C, Phillips G, Watson L, Galli L, Felix L, Edwards P, Patel V, Haines A. The effectiveness of mobile-health technologies to improve health care service delivery processes: a systematic review and meta-analysis. PLoS Med. 2013;10(1):e1001363. doi: 10.1371/journal.pmed.1001363. Epub 2013 Jan 15. PMID 23458994
- [Background] Jong S, Cuca Y, Thompson LM. Meta-analysis of Mobile Phone Reminders on HIV Patients' Retention to Care. J Mob Technol Med. 2017;6(1):5-18. doi: 10.7309/jmtm.6.1.2. PMID 30197685
- [Background] NCASC. Factsheet 1: HIV Epidemic Update of Nepal, as of December 2015. National Center for AIDS and STD Control. Kathmandu, Nepal, 2016.
- [Background] NCASC. Factsheet 6: HIV Care and Antiretroviral Therapy (ART) Services in Nepal, as of July 2016. National Center for AIDS and STD Control. Kathmandu, Nepal, 2016.
- [Background] Ayer R, Kikuchi K, Ghimire M, Shibanuma A, Pant MR, Poudel KC, Jimba M. Clinic Attendance for Antiretroviral Pills Pick-Up among HIV-Positive People in Nepal: Roles of Perceived Family Support and Associated Factors. PLoS One. 2016 Jul 20;11(7):e0159382. doi: 10.1371/journal.pone.0159382. eCollection 2016. PMID 27438024
- [Background] Kathmandu Post. Mobile subscriptions outnumber population, 2016.
- [Background] NCASC. National consolidated guidelines for treating and preventing HIV in Nepal. National Center for AIDS and STD Control. Kathmandu, Nepal, 2014.
- [Background] NCASC. National Antiretroviral Therapy Guidelines. National Center for AIDS and STD Control. Kathmandu, Nepal, 2012.
- [Background] Mugavero MJ, Davila JA, Nevin CR, Giordano TP. From access to engagement: measuring retention in outpatient HIV clinical care. AIDS Patient Care STDS. 2010 Oct;24(10):607-13. doi: 10.1089/apc.2010.0086. PMID 20858055
- [Background] Kunutsor S, Walley J, Katabira E, Muchuro S, Balidawa H, Namagala E, Ikoona E. Clinic Attendance for Medication Refills and Medication Adherence amongst an Antiretroviral Treatment Cohort in Uganda: A Prospective Study. AIDS Res Treat. 2010;2010:872396. doi: 10.1155/2010/872396. Epub 2010 Dec 19. PMID 21490907
- [Background] NCASC. National consolidated guidelines for treating and preventing HIV in Nepal. National Center for AIDS and STD Control. Kathmandu, Nepal: Ministry of health and population, 2014.
- [Background] Simbayi LC, Kalichman S, Strebel A, Cloete A, Henda N, Mqeketo A. Internalized stigma, discrimination, and depression among men and women living with HIV/AIDS in Cape Town, South Africa. Soc Sci Med. 2007 May;64(9):1823-31. doi: 10.1016/j.socscimed.2007.01.006. Epub 2007 Mar 2. PMID 17337318
- [Background] WHOQOL HIV Group. WHOQOL-HIV for quality of life assessment among people living with HIV and AIDS: results from the field test. AIDS Care. 2004 Oct;16(7):882-9. doi: 10.1080/09540120412331290194. PMID 15385243
- [Background] David J. Torgerson CJT: Designing Randomised Trials in Health, Education and the Social Sciences. New York. Palgrave Macmillan, 2008.
- [Background] Steins Bisschop CN, Courneya KS, Velthuis MJ, Monninkhof EM, Jones LW, Friedenreich C, van der Wall E, Peeters PH, May AM. Control group design, contamination and drop-out in exercise oncology trials: a systematic review. PLoS One. 2015 Mar 27;10(3):e0120996. doi: 10.1371/journal.pone.0120996. eCollection 2015. PMID 25815479
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730